CLINICAL TRIAL: NCT05926895
Title: Investigation of the Effect of Central Sensitization on Steroid Injection Response in Patients With Shoulder Pain Secondary to Rotator Cuff Lesion
Brief Title: Investigation of the Effect of Central Sensitization (CS) on Steroid Injection Response in Rotator Cuff Lesion
Acronym: CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-20
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Central Sensitisation; Subacromial Impingement Syndrome
Keywords: central sensitisation; central sensitization inventory; subacromial impingement; shoulder pain; steroid injection
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — betamethasone sodium phosphate; betamethasone dipropionate, betamethasone sodium phosphate drug combination; Prilocaine

STUDY DESIGN:
Intervention Model Description: Patients will be followed up in two groups according to the presence of central sensitization before treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with subacromial impingement syndrome (central sensitization positive) (Experimental): Subacromial steroid injection While the patient is in a sitting position the subacromial space and the rotator cuff will be evaluated with the sonosite-m turbo ultrasonography device linear probe. The area where the rotator cuff and subacromial bursa are most prominent will be determined under the deltoid muscle. The injection site is first covered with povidone iodine and then with 80% alcohol solution will be wiped to provide antisepsis. The subacromial bursa between the deltoid muscle and the rotator cuff will be advanced from lateral to medial with an inplane approach with a 21 g 38 mm needle under the guidance of ultrasonography. Bleeding after making sure that the needle tip is in the bursa by checking, 1 cc betamethasone dipropionate + betamethasone sodium phosphate and 4 cc 2% prilocaine mixture will be injected, showing that it is evenly distributed in the bursa.
  Interventions: Drug: Injection of 1 CC Betamethasone Dipropionate + Betamethasone Sodium Phosphate (Diprospan) and 4 cc 2% Prilocaine (Priloc)mixture into the subacromial space
- Patients with subacromial impingement syndrome (central sensitization negative) (Experimental): Subacromial steroid injection While the patient is in a sitting position the subacromial space and the rotator cuff will be evaluated with the sonosite-m turbo ultrasonography device linear probe. The area where the rotator cuff and subacromial bursa are most prominent will be determined under the deltoid muscle. The injection site is first covered with povidone iodine and then with 80% alcohol solution will be wiped to provide antisepsis. The subacromial bursa between the deltoid muscle and the rotator cuff will be advanced from lateral to medial with an inplane approach with a 21 g 38 mm needle under the guidance of ultrasonography. Bleeding after making sure that the needle tip is in the bursa by checking, 1 cc betamethasone dipropionate + betamethasone sodium phosphate and 4 cc 2% prilocaine mixture will be injected, showing that it is evenly distributed in the bursa.
  Interventions: Drug: Injection of 1 CC Betamethasone Dipropionate + Betamethasone Sodium Phosphate (Diprospan) and 4 cc 2% Prilocaine (Priloc)mixture into the subacromial space

INTERVENTIONS:
Drug: Injection of 1 CC Betamethasone Dipropionate + Betamethasone Sodium Phosphate (Diprospan) and 4 cc 2% Prilocaine (Priloc)mixture into the subacromial space — Treatment method used in the treatment of subacromial impingement syndrome

SUMMARY:
The goal of this clinical trial is to learn whether pretreatment central sensitization presence affect shoulder steroid injection resuls in patients with rotator cuff pathology.

The main questions it aims to answer are:

1. Is central sensitization associated with decreased treatment response?
2. Do the clinical features of patients with central sensitization differ from those of those without? Participants will be applied a shoulder injection and the treatment response will be monitored.

DETAILED DESCRIPTION:
Shoulder pain is one of the most common musculoskeletal complaints and its prevalence varies between 7-26%. One of the most common sources of pain in these patients is subacromial impingement syndrome leading to rotator cuff pathology. In patients with shoulder pain, one of the factors associated with the persistence of pain in different etiologies, especially subacromial impingement syndrome, is reported as central sensitization (CS). CS can be summarized as an increase in the response of neurons located in the central nervous system to sub-threshold stimuli. In a meta-analysis of patients with shoulder pain, a decrease in pressure pain threshold was found in 29-77% of patients, and CS in 11-24%. There is increasing data showing that CS negatively affects response to different treatments, including surgery and injections. One of the most frequently used treatments in subacromial impingement syndrome is subacromial/intra-articular shoulder injection. Although various factors have been identified in the prediction of shoulder injection results, the effect of pain sensitization on these procedures is unknown. In this study, it is planned to investigate the effect of the presence and severity of pretreatment central sensitization on the results of the shoulder injection in patients with a rotator cuff lesion or subacromial impingement.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff pathology confirmed clinically and radiologically (USG/MRI)
* Failure to respond to medical/physical treatment
* Agree to participate in the study

Exclusion Criteria:

* Shoulder trauma and history of previous shoulder surgery
* History of injection to the painful shoulder in the last 3 months
* Use of centrally acting drugs (antidepressants, pregabalin, gabapentin and myorelaxant etc.)
* History of active cancer, systemic inflammatory disease, and infection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 1 week
  The visual analog scale (VAS) is a validated subjective measure for pain, scored in the 0-10 range (0:no pain; 10: worst pain).
Visual analog scale | 1 months
  The visual analog scale (VAS) is a validated subjective measure for pain, scored in the 0-10 range (0:no pain; 10: worst pain).
Visual analog scale | 3 months
  The visual analog scale (VAS) is a validated subjective measure for pain, scored in the 0-10 range (0:no pain; 10: worst pain).
Shoulder range of motion | 1 weeks
  Goniometric measurement of flexion, extension, abduction, adduction and internal and external rotation angles of the shoulder complex
Shoulder range of motion | 1 months
  Goniometric measurement of flexion, extension, abduction, adduction and internal and external rotation angles of the shoulder complex
Shoulder range of motion | 3 months
  Goniometric measurement of flexion, extension, abduction, adduction and internal and external rotation angles of the shoulder complex

SECONDARY OUTCOMES:
QuickDASH | 1 weeks
  QuickDASH is a shortened version of the original DASH outcome measure used in upper extremity musculoskeletal disorders. Higher scores are associated with increased disability.
QuickDASH | 1 months
  QuickDASH is a shortened version of the original DASH outcome measure used in upper extremity musculoskeletal disorders. Higher scores are associated with increased disability.
QuickDASH | 3 months
  QuickDASH is a shortened version of the original DASH outcome measure used in upper extremity musculoskeletal disorders. Higher scores are associated with increased disability.
SF-36 (Short form-36) | 1 week
  The 36-item Short Form Questionnaire (SF-36) is used for objective measurement of quality of life. It consists of 8 dimensions scored between 0-100, and low scores are associated with poor in quality of life.
SF-36 (Short form-36) | 1 months
  The 36-item Short Form Questionnaire (SF-36) is used for objective measurement of quality of life. It consists of 8 dimensions scored between 0-100, and low scores are associated with poor in quality of life.
SF-36 (Short form-36) | 3 months
  The 36-item Short Form Questionnaire (SF-36) is used for objective measurement of quality of life. It consists of 8 dimensions scored between 0-100, and low scores are associated with poor in quality of life.
Hospital anxiety and depression scale (HADS) | 1 week
  Self-test questionnaire for anxiety and depression. The score between 0 and 21 for either anxiety or depression. A score of 8 and above is significant for the diagnosis of anxiety or depression.
Hospital anxiety and depression scale (HADS) | 1 month
  Self-test questionnaire for anxiety and depression. The score between 0 and 21 for either anxiety or depression. A score of 8 and above is significant for the diagnosis of anxiety or depression.
Hospital anxiety and depression scale (HADS) | 3 month
  Self-test questionnaire for anxiety and depression. The score between 0 and 21 for either anxiety or depression. A score of 8 and above is significant for the diagnosis of anxiety or depression.
hand grip strength | 1 week
  Grip strength is a measure of muscle strength or the maximum force/tension produced by one's forearm muscles and is measured with a hand dynamometer.
hand grip strength | 1 months
  Grip strength is a measure of muscle strength or the maximum force/tension produced by one's forearm muscles and is measured with a hand dynamometer.
hand grip strength | 3 months
  Grip strength is a measure of muscle strength or the maximum force/tension produced by one's forearm muscles and is measured with a hand dynamometer.
Pressure pain threshold (PPT) | 1 week
  Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. Algometer is used in the measurement and low values are interpreted in favor of increased sensitivity.
Pressure pain threshold (PPT) | 1 months
  Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. Algometer is used in the measurement and low values are interpreted in favor of increased sensitivity.
Pressure pain threshold (PPT) | 3 months
  Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. Algometer is used in the measurement and low values are interpreted in favor of increased sensitivity.

OTHER OUTCOMES:
Central sensitization inventory (CSI) | 1week
  Clinical instrument used in the diagnosis of central sensitization. A CSI part-A score of 40 and above is significant in the diagnosis.
Central sensitization inventory (CSI) | 1 months
  Clinical instrument used in the diagnosis of central sensitization. A CSI part-A score of 40 and above is significant in the diagnosis.
Central sensitization inventory (CSI) | 3 months
  Clinical scale used in the diagnosis of central sensitization. A CSI part-A score of 40 and above is significant in the diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Asst.Prof, Study Chair — Sultan Abdülhamid Han Research and Training Hospital
Locations (1):
- Sultan Abdülhamid Han Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Result] Sanchis MN, Lluch E, Nijs J, Struyf F, Kangasperko M. The role of central sensitization in shoulder pain: A systematic literature review. Semin Arthritis Rheum. 2015 Jun;44(6):710-6. doi: 10.1016/j.semarthrit.2014.11.002. Epub 2014 Nov 13. PMID 25523242
- [Result] Coronado RA, Simon CB, Valencia C, George SZ. Experimental pain responses support peripheral and central sensitization in patients with unilateral shoulder pain. Clin J Pain. 2014 Feb;30(2):143-51. doi: 10.1097/AJP.0b013e318287a2a4. PMID 23619203
- [Result] Previtali D, Bordoni V, Filardo G, Marchettini P, Guerra E, Candrian C. High Rate of Pain Sensitization in Musculoskeletal Shoulder Diseases: A Systematic Review and Meta-analysis. Clin J Pain. 2021 Mar 1;37(3):237-248. doi: 10.1097/AJP.0000000000000914. PMID 33399396
- [Result] Walankar PP, Panhale VP, Patil MM. Psychosocial factors, disability and quality of life in chronic shoulder pain patients with central sensitization. Health Psychol Res. 2020 Oct 1;8(2):8874. doi: 10.4081/hpr.2020.8874. eCollection 2020 Oct 5. PMID 33123644